CLINICAL TRIAL: NCT06119529
Title: A Phase 1, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Single-Ascending Dose Study of LY3872386 in Healthy Participants, a Multiple-Ascending Dose Study of LY3872386 in Patients With Atopic Dermatitis, and an Open-Label Multiple-Dose Evaluation of the Safety and Tolerability of Prednisone in Healthy Participants.
Brief Title: A Study of LY3872386 in Healthy Participants and Participants With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on emerging nonclinical data, the study was terminated.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18607; J4L-MC-KMAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A, B are double blind and part C is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: LY3872386 (Experimental): Single doses of LY3872386 (low dose, mid dose, and high dose) administered intravenously (IV) in healthy participants.
  Interventions: Drug: LY3872386
- Part B: LY3872386 (Experimental): Part B was planned but not initiated as study terminated early due to emerging nonclinical data.
  Interventions: Drug: LY3872386
- Part C: Prednisone (Experimental): Part C was planned but not initiated as study terminated early due to emerging nonclinical data.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Placebo administered IV in healthy participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3872386 — Administered IV.
  Arms: Part A: LY3872386; Part B: LY3872386
Drug: Prednisone — Administered orally.
  Arms: Part C: Prednisone
Drug: Placebo — Administered IV.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3872386 in healthy participants and participants with atopic dermatitis. The safety of prednisone is also evaluated in healthy participants. Blood tests will be performed to investigate how the body processes the LY3872386 following single and multiple dosing in healthy participants and participants with atopic dermatitis. Blood tests will also be performed to investigate how the body processes the prednisone in healthy participants. The study is conducted in three parts (part A, B and C). The study will last up to approximately 85, 183 and 44 days for parts A, B, and C, respectively.

ELIGIBILITY:
Inclusion Criteria:

Part A and C:

* Overtly healthy as determined by medical evaluation

  1. To qualify as Japanese for the purpose of this study, the participant must be first generation Japanese, defined as the participant's biological parents and all of the participant's biological grandparents must be of exclusive Japanese descent, and must have been born in Japan
  2. To qualify as Chinese for the purpose of this study, the participant must be, at a minimum, third-generation Chinese, defined as all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China
* Have a body mass index of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male participants who agree to use highly effective or effective methods of contraception and women not of childbearing potential may participate in part A and C

Part B:

* Participants who have a diagnosis of atopic dermatitis at least 12 months prior to screening as defined by the American Academy of Dermatology
* Have a history, documented by a physician and/or investigator, of inadequate response to existing topical medications within 6 months preceding screening, or participants who failed systemic therapies intended to treat atopic dermatitis or a history of intolerance to topical therapy
* Have a body mass index of 18.0 to 38.0 kilograms per square meter (kg/m²), inclusive
* Male participants who agree to use highly effective or effective methods of contraception, women not of childbearing potential and women of childbearing potential may participate in part B

Exclusion Criteria:

* Women who are pregnant and/or lactating
* Participants who have received live vaccine(s) (including attenuated live vaccines) or Bacillus Calmette- Guérin within 35 days of screening
* Have a history or presence of multiple or severe allergies or an anaphylactic reaction to prescription or nonprescription drugs
* Have a known history of diabetes
* Have fasting glucose level of ≥126 milligrams per deciliter (mg/dL) and glycated hemoglobin ≥6.5 percent (%) and/or taking anti-diabetes medications at screening
* Have known history of osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - CenExel ACT, Anaheim, California
  - Fortrea Clinical Research Unit, Daytona Beach, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was designed to include three parts (A, B, and C). Results are reported only for Part A, as Parts B and C were not initiated and the study was terminated early due to emerging nonclinical data.
  In Part A, single-ascending dose (SAD), of the LY3872386 (SAD Cohorts 1 and 2 and the sentinel pair in SAD Cohort 3,) was administered to healthy participants on Day 1, followed by a 12-week follow-up period.
Groups:
- Part A: Low Dose LY3872386: Participants received a single low dose of LY3872386 administered IV in healthy participants.
- Part A: Mid-dose LY3872386: Participants received a single mid-dose of LY3872386 administered IV in healthy participants.
- Part A: High Dose LY3872386: Participants received a single high dose of LY3872386 administered IV in healthy participants.
- Part A: Placebo: Participants received placebo administered IV in healthy participants.
Period: Overall Study
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part A: Placebo
Started | 6 | 6 | 1 | 5
Received at Least One Dose of Study Drug | 6 | 6 | 1 | 5
Completed | 6 | 6 | 1 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Part A: Placebo: Placebo administered IV in healthy participants.
- Total: Total of all reporting groups
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part A: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 1 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 1 | 5 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 2 | 7
  Male | 4 | 3 | 1 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 5
  Not Hispanic or Latino | 5 | 4 | 0 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 0 | 3
  White | 2 | 4 | 1 | 5 | 12
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 1 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs), Serious Adverse Event(s) (SAEs) and Other Non-serious Adverse Events (AEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality is located in the Reported Adverse Event module. Drug related TEAEs are any untoward medical occurrences that either occurs postdose or presents prior to dosing yet becomes more severe postdose, and in the opinion of the investigator is possibly related to study drug.
Time Frame: Baseline through Day 85
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Part A: Placebo IV: Placebo administered IV in healthy participants.
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part A: Placebo IV
Number analyzed (Participants) | 6 | 6 | 1 | 5
participants
  TEAEs | 0 | 2 | 0 | 0
  SAEs | 0 | 0 | 0 | 0
  AEs | 0 | 2 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With One or More TEAEs, SAEs and Other Non-serious AEs Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality is located in the Reported Adverse Event module. Drug related TEAEs are any untoward medical occurrences that either occurs postdose or presents prior to dosing yet becomes more severe postdose, and in the opinion of the investigator is possibly related to study drug. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline through Day 183
Population: Zero participants were analyzed for this outcome. Data were not captured as study was terminated early, and no participant were enrolled into Part B.
Arm/Group | Part B: LY3872386
Number analyzed (Participants) | 0

3. Primary Outcome: Part C: Number of Participants With One or More TEAEs, SAEs and Other Non-serious AEs Considered by the Investigator to be Related to Study Drug Administration
Description: as for outcome 2
Time Frame: Baseline through Day 44
Population: Zero participants were analyzed for this outcome. Data were not captured as study was terminated early, and no participant were enrolled into Part C.
Arm/Group | Part C: Prednisone
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacokinetics (PK): Part A and B: Maximum Observed Concentration (Cmax) of LY3872386
Description: Cmax of LY3872386 is reported.
Time Frame: Day 1: predose, end of infusion, 3 hours, 6 hours, and 12 hours postdose, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose (Part A)
Population: All enrolled participants who received at least one dose of LY3872386 and had evaluable PK data in Part A. Zero participants were analyzed for Part B. Data were not captured as study was terminated early, and no participant were enrolled into Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part B: LY3872386
Number analyzed (Participants) | 6 | 6 | 1 | 0
micrograms per milliliter (µg/mL) | 2.54 (16.9) | 7.89 (16.3) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 23.09 µg/mL |

5. Secondary Outcome: PK: Part A and B: Area Under the Concentration Versus Time Curve (AUC) of LY3872386
Description: Area Under the Concentration Versus Time Curve from Time Zero to tlast (AUC[0-tlast]) and Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of LY3872386 is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(µg*hr/mL)
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part B: LY3872386
Number analyzed (Participants) | 6 | 6 | 1 | 0
microgram*hour per milliliter(µg*hr/mL)
  AUC(0-tlast) of LY3872386 | 55.7 (15.6) | 328 (19.7) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 1480 µg*h/mL |
  AUC(0-∞) of LY3872386 | 65.8 (18.6) | 337 (20.3) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 1560 µg*h/mL |

6. Secondary Outcome: PK: Part C: Cmax of Prednisone and Prednisolone
Description: Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Predose up to 12 hours post dose on day 14 and day 30
Population: as for outcome 3
Arm/Group | Part C: Prednisone
Number analyzed (Participants) | 0

7. Secondary Outcome: PK: Part C: AUC of Prednisone and Prednisolone
Description: Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Predose up to 12 hours post dose on day 14 and day 30
Population: as for outcome 3
Arm/Group | Part C: Prednisone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 85
Description: All randomized participants who received at least one dose of the study drug.
Arm/Group | Part A: Low Dose LY3872386 | Part A: Mid-dose LY3872386 | Part A: High Dose LY3872386 | Part A: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 0/1 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Low Dose LY3872386 (N=6) | Part A: Mid-dose LY3872386 (N=6) | Part A: High Dose LY3872386 (N=1) | Part A: Placebo (N=5)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on the emerging nonclinical data, Study KMAA was terminated after the dosing of participants in SAD Cohorts 1 and 2 (Dose 1 IV and Dose 2 IV) and the sentinel pair in SAD Cohort 3 (Dose 3 IV).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT06119529/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT06119529/SAP_001.pdf